CLINICAL TRIAL: NCT03444662
Title: The Combination of Citicoline and Omega-3 on Attention in Healthy Subjects
Brief Title: The Combination Effect of Citicoline and Omega-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyowa Hakko Bio Co., Ltd. (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16518
Record Dates: First submitted 2018-02-14; First posted 2018-02-23 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Cytidine Diphosphate Choline; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Intervention: Dietary Supplement: Placebo supplement
  Interventions: Dietary Supplement: Placebo supplement
- Cognizin and Omega-3 (Experimental): Intervention: Dietary Supplement: Citicoline and Omega-3 supplement
  Interventions: Dietary Supplement: Citicoline and Omega-3 supplement
- Omega-3 (Experimental): Intervention: Dietary Supplement: Omega-3 supplement
  Interventions: Dietary Supplement: Omega-3 supplement

INTERVENTIONS:
Dietary Supplement: Placebo supplement — Cellulose and Sunflower oil
  Other Names: Placebo
  Arms: Placebo
Dietary Supplement: Citicoline and Omega-3 supplement — Citicoline and Omega-3
  Other Names: Cognizin and Omega-3
  Arms: Cognizin and Omega-3
Dietary Supplement: Omega-3 supplement — Cellulose and Omega-3
  Other Names: Omega-3
  Arms: Omega-3

SUMMARY:
The goal of this study is to determine the effects of Citicoline plus Omega-3 or Omega-3 alone versus placebo on attention in non-demented healthy older adults.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial. The investigators hypothesize that supplementation of Citicoline plus Omega-3 will improve attention in healthy adults age 55 years and older, compared to placebo. The study is designed as 3-arm, parallel group study comparing placebo, Omega-3 only, and Citicoline plus Omega-3.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* If female, must be post-menopausal
* Non-demented
* Not depressed
* General health status that will not interfere with the participant's ability to complete the study
* No history of neurological disorder
* Screening laboratory values within normal limits or, if abnormal, deemed clinically insignificant by the investigator
* Sufficient English language skills to complete all testing

Exclusion Criteria:

* Alzheimer's, Dementia or other neurological disease
* Fish intake of 6 ounce serving once a week 3 months prior to enrollment; Omega-3 supplement intake (e.g. fish oil capsules, cod liver oil, or flaxseed oil) less than 3 months prior to enrollment.
* Citicoline supplementation 3 months prior to enrollment
* Prescriptions medications:

  1. Anticoagulation therapy: Vitamin K antagonist: warfarin (Coumadin, jantoven), Factor Xa inhibitors: rivaroxaban (xarelto), fondaparinux (arixtra), dibigatran (pradaxa), apixaban (eliquis); Low molecular weight heparins: dalteparin (fragmin), enoxaparin (lovenox)
  2. Dementia medications (e.g. anticholinesterase inhibitors, memantine)
  3. Diagnosis of Adult Attention Deficit Disorder (ADD) or Attention Deficit Hyperactivity Disorder (ADHD) and/or taking stimulants (e.g. dextroamphetamine sulfate, methylphenidate HCL, dextroamphetamine Sulf-Saccharate)
* Body Mass Index > 30
* Enrollment in another treatment study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Accuracy (percent correct) on an attention task (Conners continuous performance test3) | 16 weeks

SECONDARY OUTCOMES:
Scores of Neuropsychological test battery from the Uniform Data Set | 16 weeks

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as monitored by recording a comprehensive metabolic panel, complete blood count and prothrombin time-international normalized ratio | 16 weeks
Plasma fatty acid levels | 16 weeks
Apolipoprotein E genotype | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States